CLINICAL TRIAL: NCT06303284
Title: Post-surgical Outcomes With Anabolic Agent Use in High-risk Ankle Fractures: A Pilot RCT
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pending
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Ankle Fractures
MeSH Terms: conditions — Ankle Fractures | interventions — Teriparatide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Teriparatide (Experimental): 20 µg subcutaneous Teriparatide injection once daily for 3 months in the post-operative ankle fracture population.
  Interventions: Drug: subcutaneous Teriparatide injection
- placebo (Sham Comparator): 20 µg subcutaneous saline placebo injection once daily for 3 months in the post-operative ankle fracture population.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: subcutaneous Teriparatide injection — 20 µg subcutaneous (SC) Teriparatide injection
  Other Names: Teriparatide
  Arms: Teriparatide
Other: placebo — placebo 20 µg subcutaneous saline placebo injection once daily for 3 months in the post-operative ankle fracture population.
  Arms: placebo

SUMMARY:
As the global population ages and the prevalence of poor bone health increases among older patients with ankle fractures, so does the risk of post-surgical complications. Prevention of post-surgical complications is of paramount importance to reducing morbidity, mortality, and healthcare costs.

There is growing evidence to support the use of bone-building medications, such as Teriparatide, in patients who have delayed fracture healing or non-unions; however, these medications have yet to be investigated in elderly patients with ankle fractures at high risk for delayed fracture healing and post-operative complications. This project aims to assess the safety and efficacy of short-term Teriparatide use in improving outcomes in a population most likely to suffer post-operative complications.

The proposed study is a pilot randomized controlled trial (RCT) with patients 60 years or older with an additional risk factor for delayed healing (i.e., osteoporosis, diabetes, vascular disease) who require ankle fracture surgery. Participants will be randomized to receive the study medication (Teriparatide) or placebo for three months. The primary objective of this study is to acquire vital data (i.e., recruitment rates, follow-up rates, adherence to treatment assignment) required to determine the feasibility of a full-scale multi-centre RCT. Additional aims are to evaluate repeat surgery, complications, time-to-union, and 90-day mortality. A complete a socio-economic and feasibility analysis will be completed.

This study will evaluate the novel clinical approach of augmenting surgical fixation with a medication to build bone density and strength, thereby improving bone health, preventing complications, and improving outcomes. This study will also inform planning for a larger clinical trial to reduce the morbidity, mortality, and cost associated with complications in this high-risk population.

DETAILED DESCRIPTION:
Background: Delayed healing, implant failure, loss of reduction, and infection rates are common post-operative complications following ankle fracture fixation among patients aged 60 years or older with compromised soft tissue and/or metabolic challenges. There is growing evidence to support the safety and efficacy of using anabolic agents in achieving osseous union in the setting of delayed fracture healing and nonunion. Teriparatide has been prescribed for the treatment of osteoporosis, with very few serious adverse events reported. Therefore, the goals of the proposed research are to examine the safety and efficacy of Teriparatide use for high-risk acute ankle fractures and to determine the feasibility of a full-scale trial. This new knowledge will inform the implementation of Teriparatide for improved fracture healing.

Specific Aims (SA): The investigators hypothesize that the short-term use of the anabolic agent, Teriparatide, will augment fracture fixation and result in lower complication rates. Our specific aims include: SA1) Evaluate the feasibility of a definitive, full-scale randomized controlled trial comparing Teriparatide with a placebo; SA2) Compare the post-operative complication rate between short-term augmentation with Teriparatide and a placebo; and SA3) Evaluate the safety and efficacy of Teriparatide use.

Methods: This study is a multi-center double-blinded pilot randomized controlled trial (RCT) with patients 60 years or older with an additional risk factor for delayed healing (i.e., osteoporosis, diabetes, vascular disease) who require ankle fracture surgery. Participants will be randomized to receive the study medication (Teriparatide) or placebo for three months. The primary objective of this study is to acquire vital data (i.e., recruitment rates, follow-up rates, adherence to treatment assignment) required to determine the feasibility of a full-scale multi-center RCT. Additional aims are to evaluate repeat surgery, complications, time-to-union, and 90-day mortality. A complete a socio-economic and feasibility analysis will be completed.

Significance: Delayed healing, implant failure, loss of reduction, and infection rates continue to be devastating complications of ankle fracture fixation that profoundly impact patients and their families, surgeons, and the healthcare system. It is imperative that the investigators evaluate innovative strategies for improving outcomes for these high-risk patients. The multi-disciplinary team of investigators has designed this project to generate new knowledge about the safety and efficacy of using Teriparatide in the acute fracture setting in order to reduce complications, morbidity, and mortality in this vulnerable population. By addressing knowledge gaps and promoting evidence-based education and interventions, the project aims to have a sustainable impact on scientific knowledge, clinical practice, and ultimately, the well-being of elderly patients undergoing ankle fracture fixation.

ELIGIBILITY:
Inclusion Criteria:

* Our study will include men and women over 60 years of age presenting to the emergency department with low energy ankle fractures (fall from standing height) requiring surgical treatment and who have one or more of the following risk factors, diabetes, osteoporosis, renal disease, steroid use, smoking history, peripheral neuropathy and/or vascular disease.

Exclusion Criteria:

* Individuals will be excluded if they have received previous Teriparatide therapy, or they have hypercalcemia or hyperparathyroidism, as these are precautions to the use of Teriparatide.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Participant recruitment rate | 2 years
  Estimate of the mean monthly recruitment rate across participating sites

SECONDARY OUTCOMES:
Incidence of composite measure of complications | 3 month after surgery
  Estimate of composite measure of complication (revision surgery, infection, non-union).
Adverse events | 3 month after surgery
  Estimate of intervention related adverse events
modified Radiological Union Scale for Tibia [RUST] score), | 2 week, 4 week, 2 months, 3 months, 4 months, 5 months, 6 months post operative.
  Tool for radiographic assessment of fracture healing
Olerud Molander Score | within 48 hours of surgery, 3 month and 6 months after surgery.
  a functional rating scale from 0 (totally impaired) to 100 (completely unimpaired)
EuroQol five dimensions [EQ-5D] | within 48 hours of surgery, 3 month and 6 months after surgery.
  Quality of life measure
short form-12 [SF-12] | within 48 hours of surgery, 3 month and 6 months after surgery.
  Quality of life measure
pain visual analogue score [VAS] | within 48 hours of surgery, 3 month and 6 months after surgery.
  Pain intensity measure
time-to-fracture union | 6 month post operative
  the time between fracture and radiological healing of the fracture
90 day mortality | 3 month post operative
  Mortality rate after 90 days of the surgery
Bone mineral density | 2 week and 3 month post operative
  Bone mineral density scan
Total cost and QALYs | 3 month post operative
  Measurement of the incremental cost per QALY gained for the more effective treatment option.

IPD SHARING:
Plan to Share IPD: Undecided